CLINICAL TRIAL: NCT01322997
Title: Robotic Brace Incorporating EMG for Moderate Affected Arm Impairment After Stroke
Brief Title: Robotic Brace Incorporating Electromyography (EMG) for Moderate Affected Arm Impairment After Stroke
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Responsible Party: Stephen J. Page, PhD, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R03HD062545-01 (NIH)
Record Dates: First submitted 2011-03-16; First posted 2011-03-25 (Estimated); Last update posted 2011-03-25 (Estimated); Status verified 2011-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — N-myc downstream-regulated gene 1 protein

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Myomo + RTP (Experimental): This group will be administered a regimen comprised of repetitive task specific practice (RTP) in conjunction with use of the robotic brace described elsewhere in this record.
  Interventions: Device: Myomo e100 Robot and repetitive task specific training
- Myomo (Active Comparator): Patients in this group will only be administered the robotic brace described elsewhere in this record.
  Interventions: Device: Myomo e100 neurorobotic brace
- RTP only (Active Comparator): Patients in this group will be administered repetitive task specific practice (RTP), emphasizing use of their affected arms during performance of valued, functional tasks.
  Interventions: Behavioral: Repetitive task specific training (RTP) targeting the affected arm

INTERVENTIONS:
Device: Myomo e100 Robot and repetitive task specific training — Subjects in this group will be administered about an hour/day of therapy targeting the affected arm. This therapy will include about 1/2 an hour of use of a robot that targets arm function and assists with the movement of the affected arm, and about 1/2 an hour of repetitive task specific training (TRP) using the affected arm.
  Arms: Myomo + RTP
Behavioral: Repetitive task specific training (RTP) targeting the affected arm — Subjects in this group will be administered about an hour/day of therapy targeting the affected arm. This therapy will include consist of repetitive task specific training (RTP) using the affected arm, in which patients use the arm to relearn valued movements using their arms.
  Arms: RTP only
Device: Myomo e100 neurorobotic brace — Subjects in this group will be administered about an hour/day of therapy targeting the affected arm. Subjects will use a robot that targets arm function and assists with the movement of the affected arm.
  Arms: Myomo

SUMMARY:
Stroke is the leading cause of disability in the United States. One of the reasons that it is so disabling is because of upper extremity hemiparesis (weakness in one arm), which is commonly seen after stroke.

The objective of this research is to see if a robotic system worn on the weakened arm like a brace is more useful in improving the strength and coordination of the affected arm, and those of other stroke survivors, than therapy only. Muscle weakness and lack of coordination after a stroke have great effects on how severely disabled the arm is and on quality of life after a stroke.

In this study, patients may be administered a new robotic brace as part of treatment for their affected arms. If they use this brace, your electromyography (EMG) signals will be used to control the powered arm brace. EMG signals are the small electrical signals that result from the actions of the muscles. The system will "listen" to patients' muscles, using small sensors that sit on top of the skin. The device will give the arm a "power-assist" when patients bend or straighten their elbows. The investigators want to test how easy and effective this system is to use. The investigators hypothesize that people using the robot will be more successful in their rehabilitative efforts - and that their movement will improve more - than people receiving traditional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Upper extremity Fugl Meyer score >10-< 25
* presence of volitionally activated EMG signal from the paretic biceps brachii of at least 5 ųV in amplitude
* stroke experienced > 1 month prior to study enrollment;
* a score > 24 on the Folstein Mini Mental Status Examination (MMSE)
* age > 35 < 85
* have experienced one stroke
* discharged from all forms of physical rehabilitation
* Myomo brace fits on affected arm properly and without discomfort (i.e., no red marks or discomfort observed in 10 minutes of use during fitting).

Exclusion Criteria:

* < 35 years old
* excessive pain in the affected hand, arm or shoulder, as measured by a score > 5 on a 10-point visual analog scale
* excessive spasticity at the affected elbow, as defined as a score of > 4 on the Modified Ashworth Spasticity Scale
* currently participating in any experimental rehabilitation or drug studies
* apraxia (< 2.5 on the Alexander scale)
* severe sensory loss in affected hand (Nottingham sensory scale at least 75% of normal)
* severe language deficits (score < 2 on NIH Stroke Scale question 9)
* Stroke that occurred in the brainstem
* A current medical history of uncontrolled cardiovascular, or pulmonary disease, or other disease that would preclude involvement in a therapeutic treatment
* History of neurological disorder other than stroke (other neurological disorders may affect the upper extremity motor performance of subjects.)
* Other significant pain or skin irritation in the upper extremity that would be exacerbated if by the use of the brace
* Substantial contracture of elbow, defined as > 20 degrees of elbow flexion, as measured at the baseline evaluation.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to after intervention and 3 months after intervention in the amount of active movement at each joint of the affected arm. This will be measured using the upper extremity section of the Fugl-Meyer Assessment. | Twice before intervention; once after intervention; 2 months after intervention.
  The primary outcome in this study is arm impairment. We will measure this using the Fugl-Meyer; a stroke-specific measure that determines how much active movement patients exhibit at each joint of the affected upper extremity.

CONTACTS AND LOCATIONS:
Locations (1):
- Univcersity of Cincinnati, Cincinnati, Ohio, United States